CLINICAL TRIAL: NCT00554021
Title: Infections Associated With the Use of Central Venous Catheters Related in Critical Care Center.
Brief Title: Infections Related Central Venous Catheters
Acronym: CVL
Status: Completed | Type: Observational
Sponsor: National Defense Medical College, Japan (Other)
Responsible Party: Kahoko Nishikawa, NDMC
Other Study IDs: NDMC-CV0001
Record Dates: First submitted 2007-11-05; First posted 2007-11-06 (Estimated); Last update posted 2009-06-12 (Estimated); Status verified 2009-06

CONDITIONS: SIRS
Keywords: Central venous catheter; nosocomial infection
MeSH Terms: conditions — Cross Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We will use the DNA from the only clinical isolated bacteria.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: Department of Traumatology and Critical Care Medicine, National Defense Medical College

SUMMARY:
The purpose of this study is to clarify the relationship between SIRS (Systemic inflammatory response syndrome) and the infection associated with the use of central venous catheters at Critical Care center in National Defense Medical College, Japan.

DETAILED DESCRIPTION:
The doctor would remove the inserted catheter from the patient, if the patient shows SIRS. At the same time, the tip of used catheter and blood from the patient are checked whether the pathogenic bacteria exists or not by general bacterial protocol and blood culture test on a routine application. Unfortunately, these tests not always clarified their cause of SIRS. Therefore we conduct this investigation to establish the useful protocol for pathogenic bacteria. We check the pathogenic bacteria not only tip but through the whole catheter in Central Venous Catheter using general bacterial protocol and SEM observation. Additionally, we compared that sputum, urine, skin and blood from the patient for bacteria check.

ELIGIBILITY:
Inclusion Criteria:

* A patient has been inserted with central venous line over 24 hours.

Ages: 14 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Critical Care staff
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2007-11; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Culture of bacteria with in central venous catheter. Morbidity and mortality of a patient with multiple resistant bacteria associated with use of the catheter. | four months

CONTACTS AND LOCATIONS:
Overall Officials: Kahoko NISHIKAWA, PHD, Study Director — National Defense Medical College
Locations (1):
- Department of Traumatology and Critical Care of Medicine, Tokorozawa, Saitama, Japan